CLINICAL TRIAL: NCT05104502
Title: Immunomodulatory Effects of Fasting in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1816627
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Experimental): Dietary fasting.
  Interventions: Behavioral: Dietary Fasting

INTERVENTIONS:
Behavioral: Dietary Fasting — The study will consist of two days of eating a "controlled habitual diet" and one 36-hour period of water-only fasting with glucose monitoring as a measure of compliance. Water intake will be limited to 2 liters/day to prevent electrolyte abnormalities. Subjects will undergo 4 separate blood-draws consisting of an overnight fasted sample (Baseline), a 2-hour postprandial sample (Fed), a 36-hour fasted sample (Fasted), and final 2-hour postprandial sample after the fasting period (Refed).

SUMMARY:
This is a clinical trial assessing the effects of fasting on the immune system in healthy adults. Immune profiling, gene expression profiling, and flow cytometry on peripheral blood mononuclear cells (PBMCs) will be performed and we hypothesize that a period of fasting will alter the immune system in healthy adults.

DETAILED DESCRIPTION:
Dietary restriction (DR) is an intervention demonstrated to increase healthy lifespan in various model organisms including yeast, worms, mice, and rhesus monkeys (Lee et al., 2016, Fontana et al., 2015). It has been investigated extensively as a therapeutic modality in metabolic disease such as hypertension, cardiovascular disease, and obesity, with evidence of benefit independent of weight loss (Wilkinson et al., 2020, Zhu et al., 2020, Di Francesco et al., 2018). The major DR regimens include caloric restriction (CR) (Fontana et al., 2010), time-restricted feeding (TRF) (Brandhorst et al., 2015), fasting mimicking diets (FMD) (Mirzaei et al., 2014), and intermittent fasting (IF) (Chaix et al., 2014). Within the broader, poorly defined concept of IF, specific regimens exist that have yet to be standardized, including alternate-day fasting (ADF), 5:2 intermittent fasting (fasting 2 days per week), and daily TRF (typically restricting eating to an 8 hour window with 16 hours of fasting) (Chaix et al., 2014, Stekovic et al., 2019).

Studies of the effects of several different forms of DR on the immune system have shown both pro- and anti-inflammatory effects on immune responses, particularly with chronic calorie restriction (Choi et al., 2017). Certain periodic dietary restrictions prevent immune dysfunction and restore normal immune functioning by decreasing the number of circulating autoimmune cells from circulation and activating tissue regenerative capacity (Cheng et al., 2014). Although both chronic CR and nutrient-restricted FMD require substantial lifestyle modifications and can prove challenging in terms of adherence, forms of TRF and IF provide reasonable alternatives while showing similar efficacy. This makes forms of DR involving fasting rather than CR more appealing as a clinical intervention.

While multiple studies have shown positive effects on the immune system with various IF regimens in the setting of rheumatoid arthritis (Müller et al., 2001), multiple sclerosis, and cancer, mechanistic data in healthy humans are lacking. Recent studies have demonstrated changes in immune cell distribution with various regimens of CR and IF in murine models, supporting the exploration of potentially similar changes in healthy humans (Nagai et al. 2019). In order to study mechanistic details of the immune changes seen with DR in healthy humans, we designed this trial to examine the effects of fasting dose on multiple immune cell populations and relevant cell surface markers. While we observe a cohort over what is effectively only a single cycle of ADF, here we make an important step in characterizing the immune modulation occurring with ADF. This is one of the most studied fasting regimens, with substantial possibility for use as a clinical therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years, to constitute a young study population
* Gender: male subjects, to control for gender differences
* BMI: 19-27 kg/m2 to constitute a normal/healthy weight population
* Weight: 120 lbs or more
* Fasting glucose: 70-100 mg/dL, to ensure that fasting can be tolerated without inducing dangerously low levels of blood glucose
* Subjects must be willing to undergo a period of 36 hours of water-only fasting
* Subjects must be willing to collect samples of each bowel movement produced throughout the entire study period for microbiome analysis
* Subjects must be willing to collect blood pricks for blood glucose levels using a Contour Next One Blood Glucose Testing Kit during the fasting stage of the study protocol.

Exclusion Criteria:

* Current smoking
* Anemia
* Pregnancy or current breastfeeding
* Chronic diseases including diabetes mellitus, thyroid disease, metabolic syndrome, cancer, or previous cardiovascular events
* Gastrointestinal diseases including irritable bowel syndrome, Crohn's disease, ulcerative colitis, celiac disease
* Consumption of >1 alcoholic drink/day
* Extreme dietary or exercise patterns
* Recent weight fluctuations (greater than 10% in the last six months)
* Regular use of over-the-counter allergy or pain medications (>1/week)
* Taking prescription lipid medications (e.g. statins) or other supplements known to alter lipoprotein metabolism such as isoflavones
* Use of hormonal birth control including oral contraception pills, hormonal IUDs or rings, or hormonal birth control patches

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in peripheral blood mononuclear cells | 7 months
  Changes in surface proteins and glycoproteins of peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States